CLINICAL TRIAL: NCT01227096
Title: National Natural Science Foundation of China
Brief Title: Randomized Controlled Trial of the Effects of Electroacupuncture Preconditioning in Children Undergoing Cardiac Surgery
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Air Force Military Medical University, China (Other)
Collaborators: National Natural Science Foundation of China (Other Government)
Responsible Party: Xiong Li-Ze, Xijing Hospital of Fourth Military Medical University
Other Study IDs: NSFC3090091-6
Record Dates: First submitted 2010-10-22; First posted 2010-10-25 (Estimated); Last update posted 2011-06-23 (Estimated); Status verified 2010-10

CONDITIONS: Congenital Heart Defects
Keywords: electroacupuncture pediatric cardioprotection
MeSH Terms: conditions — Heart Defects, Congenital

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Biospecimen Retention: Samples Without DNA — blood serum
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- Electro-acupuncture, Control
  Interventions: Device: Electrical acupuncture stimulation
- Preconditioning, No preconditioning

INTERVENTIONS:
Device: Electrical acupuncture stimulation — electroacupuncture would be administered on the bilateral P6 acupoint after anesthesia induction, but prior to surgery.
  Other Names: Suzhou Hua Tuo Medical Instruments Co, Ltd, Suzhou, China
  Groups: Electro-acupuncture, Control

SUMMARY:
The purpose of this study is to determine whether electroacupuncture preconditioning would provide protection against myocardial Ischemic-Reperfusion injury and systemic inflammation in children undergoing CPB for repair of congenital heart defects.

DETAILED DESCRIPTION:
2-12 years old children undergoing repair of congenital heart defects were included, except for those with server pulmonary arterial hypertension, chromosomal defects, airway and parenchymal lung disease, immunodeficiency, or blood disorders were excluded. Children were equal randomized to EAPC(electroacupuncture preconditioning)or control group. Electroacupuncture was administered on the bilateral P6 acupoint after anesthesia induction, but prior to surgery in EAPC group. Control patients underwent sham placement of the electrode the arm without stimulation. The duration of cardiopulmonary bypass and aortic cross-clamp time was recorded. Myocardial injury was assessed by cardiac heart-type fatty acid-binding protein (HFAP) and cardiac troponin I (cTnI>0.40 ng/mL). 8-isoprostane , C-reactive protein, cytokines were measured pre- and postoperatively.

ELIGIBILITY:
Inclusion Criteria:

* Aged 2-12 years children undergoing repair of congenital heart defects without server pulmonary arterial hypertension or systematic disease.
* Get an informed consent from parental.

Exclusion Criteria:

* Patient's age is less than 2 years or more than 12 years.
* Patient with isolated atrial septal defect undergoing repair via thoracoscope completion.
* Patients with chromosomal defects, airway and parenchymal lung disease, immunodeficiency, or blood disorders.
* Patients without an informed consent from parental.

Ages: 2 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: 2-12 years old children undergoing all types of open-heart surgery were included.
Sampling Method: Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2010-10; Primary Completion 2011-05 (Actual); Study Completion 2011-07 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Xin-Li Ni, PhD, Principal Investigator — Department of Anesthesiology of Xijing Hospital; Li-Ze Xiong, PhD, Study Chair — Xijing Hospital of Fouth Military Medical University; Qiang Wang, PhD, Study Director — Department of Anesthesiology of Xijing Hospital
Locations (1):
- Xijing Hospital, Xi’an, Shanxi, China